CLINICAL TRIAL: NCT06052826
Title: Geriatric (G) Assessment Guided Optimization (O) to Accelerate Functional Recovery After Chimeric Antigen Receptor T-Cell (CAR-T) Therapy for Patients 60 Years and Older With B-Cell Non-Hodgkin Lymphoma or Multiple Myeloma (GOCART)
Brief Title: Geriatric Assessment Guided Interventions to Accelerate Functional Recovery After CAR-T Therapy for Patients 60 Years and Older With B-cell Non-Hodgkin Lymphoma or Multiple Myeloma, GOCART Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22422; NCI-2023-04359 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22422 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-09-11; First posted 2023-09-25 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: B-Cell Non-Hodgkin Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Lymphoma, B-Cell; Multiple Myeloma | interventions — Practice Guidelines as Topic; Standard of Care; Geriatric Assessment; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (PT, cognitive education, nutrition education) (Experimental): Patients undergo GA before lymphodepleting chemotherapy and recommendations based on assessment results communicated to treating physicians. Patients receive PT and delirium prevention education prior to lymphodepletion, at least once before CAR-T therapy, at least 2 times a week while inpatient, and at least once every other week outpatient up to day 30. Additionally, patients receive personalized nutritional guidance from a registered dietician prior to lymphodepletion, prior to CAR-T therapy and at least once a week up to day 30.
  Interventions: Other: Cognitive Intervention; Other: Comprehensive Geriatric Assessment; Other: Nutritional Intervention; Procedure: Physical Therapy; Other: Questionnaire Administration
- Arm II (standard of care) (Active Comparator): Patients undergo GA and receive standard of care throughout study.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Undergo standard of care
  Other Names: standard of care; standard therapy
  Arms: Arm II (standard of care)
Other: Cognitive Intervention — Receive delirium prevention education
  Arms: Arm I (PT, cognitive education, nutrition education)
Other: Comprehensive Geriatric Assessment — Undergo geriatric assessment
  Arms: Arm I (PT, cognitive education, nutrition education)
Other: Nutritional Intervention — Undergo nutritional optimization
  Arms: Arm I (PT, cognitive education, nutrition education)
Procedure: Physical Therapy — Undergo physical function optimization
  Other Names: Physiatric Procedure; Physical Medicine Procedure; Physical Therapeutics; Physical Therapy Procedure; Physiotherapy; Physiotherapy Procedure; PT
  Arms: Arm I (PT, cognitive education, nutrition education)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial compares the effectiveness of geriatric assessment (GA) guided interventions to accelerate functional recovery after chimeric antigen receptor T-cell (CAR-T) therapy compared to standard of care (SOC) in patients 60 years and older with B-cell non-Hodgkin lymphoma (NHL) or multiple myeloma (MM). A large number of patients diagnosed with cancer are over the age of 60, yet most cancer treatments are developed for younger patients. Therefore, older patients may be less likely to be offered stronger treatments, such as CAR-T therapy, due to possible side effects. Geriatric assessment is a multi-dimensional health assessment tool combining patient reported and objective measures covering physical function, mental processes (cognitive), and nutrition. Pre-treatment assessments may identify weaknesses in older adults and may guide interventions for physical therapy, cognitive changes and nutrition to decrease CAR-T therapy side effects and improve care in older adults with NHL or MM.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the effects of a GA-informed multi-disciplinary intervention in attenuating physical function decline among older patients receiving CAR-T therapy at day +30 post-CAR-T infusion.

SECONDARY OBJECTIVES:

I. Determine success in coordinating trimodality optimization before lymphodepletion.

II. Compare rates of geriatric syndromes of frailty, cognitive impairment and malnourishment in SOC and GA-intervention cohorts at 30 days post-CAR-T infusion.

III. Evaluate rates and duration of CAR-T related neurotoxicity in SOC and GA-intervention groups.

EXPLORATORY OBJECTIVES:

I. Quantify trimodality optimization intensity throughout treatment course. II. Compare longitudinal trajectory of Short Physical Performance Battery (SPPB), frailty, cognitive impairment and malnourishment between the two arms, at day +100 post-CAR-T infusion.

III. Evaluate quality of life trajectories using the Patient Reported Outcomes Measurement Information System (PROMIS) Global Health Scale at baseline and days +30 and +100 in both cohorts.

IV. Incidence of intensive care unit (ICU) admissions by day 100. V. Overall survival, response rate and progression-free survival through one year.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo GA before lymphodepleting chemotherapy and recommendations based on assessment results communicated to treating physicians. Patients receive physical therapy (PT) and delirium prevention education prior to lymphodepletion, at least once before CAR-T therapy, at least 2 times a week while inpatient, and at least once every other week outpatient up to day 30. Additionally, patients receive personalized nutritional guidance from a registered dietician prior to lymphodepletion, prior to CAR-T therapy and at least once a week up to day 30.

ARM II: Patients undergo GA and receive standard of care throughout study.

After completion of study treatment, patients are followed up at day 100 and then up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Patient's physician must agree for patient participation. A physician may elect to provide blanket agreement for participation of any eligible CAR-T patient under their care
* Ability to read English, or Spanish. Other languages will be acceptable with site principal investigator (PI) agreement if surveys are available and language does not preclude completing study procedures
* Age: >= 60 years at the time of enrollment
* Scheduled to receive an Food and Drug Administration (FDA)-approved CAR-T for treatment of multiple myeloma or B-cell non- Hodgkin lymphoma
* Willing and able to complete study requirements
* Patients expect to be able to participate at least once before lymphodepletion with trimodality optimization visits

Exclusion Criteria:

* Prior CAR-T therapy
* Any condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2026-10-05 (Estimated); Study Completion 2026-10-05 (Estimated)

PRIMARY OUTCOMES:
Changes in Short Physical Performance Battery (SPPB) | From baseline to day 30 after chimeric antigen receptor T-cell (CAR-T) infusion
  T-test will be used to compare SPPB changes score between two arms at 30 days after CAR-T infusion.

SECONDARY OUTCOMES:
Successful in coordinating initial optimization | From enrollment to start of lymphodepletion
  A physical or virtual visit will be tabulated separately for functional optimization, delirium prevention and nutrition. Adherence will be deemed to have been met if >=70% or more comlete tri-modality optimization before lymphodepletion in the modified intent to treat population.
Frailty progression | At 30 days post CAR-T infusion
  Frailty progression will be defined as a score of 3 or more at T2 if T1 not frail (<3); if frail at T1 (score 3-5), any worsening of the score; a score of 5 at day 30 if baseline score already at the maximum frailty of 5.
Cognitive impairment | At 30 days post CAR-T infusion
  Assessed using the Montreal Cognitive Assessment (MoCA). Cognitive impairment defined as MoCA score of < 23 or unable to complete the MoCA due to cognitive impairment. The proportion of patients with cognitive impairment at day 30, irrespective of baseline cognition, will be compared between the two arms using Chi-square test.
Weight loss | Up to 30 days post CAR-T infusion
  Malnourishment will be measured using weight loss and dichotomized as > 5% weight loss from baseline to day +30. The proportion of patients with over 5% weight loss from T1 to T2 will be compared between the two arms using Chi-square test.
CAR-T associated neurotoxicity | Up to day 100
  Assessed using American Society for Transplantation and Cellular Therapy consensus grading for cytokine release syndrome and immune effector cell-associated neurotoxicity syndrome (ICANS). The time to neurotoxicity (days), the maximum grade (1-4) and the duration of neurotoxicity (days) will be recorded. The cumulative incidence of ICANS (percentages) will be compared between arms as well as the maximum grade (1-4), and duration of neurotoxicity (days).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Artz, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States